CLINICAL TRIAL: NCT02240368
Title: Performance Evaluation of the Depth of Anesthesia Monitors in Pediatric Surgery. Bispectral VISTA and ENTROPY Monitor for Pediatric Anesthesia.
Brief Title: Performance Evaluation of the Depth of Anesthesia Monitors in Pediatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Alberto Sciusco, Medical doctor, University of Foggia
Other Study IDs: A01
Record Dates: First submitted 2014-08-31; First posted 2014-09-15 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia; Child
Keywords: Depth anesthesia monitors; Children anesthesia; Bispectral monitor; Entropy monitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: Children age between 1 month to 12 months
- Group 2: Children age between 13 months and 36 months
- Group 3: Children age between 37 months to 144 months

SUMMARY:
The purpose of this study is to determine how Bispectral index (BIS) and Entropy EEG monitors agree between themselves and with end-tidal concentration of sevoflurane (ETsevo) in relationship with the age in the pediatric surgery setting.

Bispectral index (BIS) and Entropy EEG monitors performance and utility is well established in adult general anesthesia.

Their utility is yet undefined in the pediatric population as age seems to affect their ability to track the cerebral hypnotic state in children.

DETAILED DESCRIPTION:
All patients monitored applying standard device for blood pressure, electrocardiogram and pulse oximeter for routine monitor of anesthesia in pediatric surgery. Bispectral VISTA monitor and Entropy monitor applied for monitoring the depth of anesthesia. The investigators will not assign any specific interventions to the subjects of the study.

ELIGIBILITY:
Inclusion Criteria:

* physical status classification (ASA) I - II
* general balanced anesthesia
* mechanically ventilated with laryngeal mask

Exclusion Criteria:

* severe developmental delay
* neurological disorders or receiving treatment with antiepileptic or stimulant
* patients with preexisting lung or cardiac disease
* airway abnormalities
* marked skin sensitivity and conditions where the placement of the BIS and Entropy sensor or process of assessment would interfere with the surgery procedure.
* patients receiving local anaesthesia, regional block combined with general anaesthesia
* sedation administered by non anesthesiologists for invasive and noninvasive diagnostic or therapeutic procedures

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with age ≤ 12 years old scheduled to undergo general anesthesia and mechanical ventilation for elective surgery
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Dambrosio, Medic, Study Chair — University of Foggia; Gilda Cinnella, Medic, Study Director — University of Foggia; Alberto Sciusco, medic, Principal Investigator — University of Foggia; Pasquale Raimondo, Medic, Principal Investigator — University of Foggia
Locations (1):
- Ospedali Riuniti, Foggia, FG, Italy

REFERENCES:
- See also: Speciality school of anesthesia of University of Foggia — http://www.anestesia.unifg.it/
- See also: University of Foggia — http://www.unifg.it/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 9 | 22 | 19
Completed | 8 | 22 | 18
Not Completed | 1 | 0 | 1
Not completed — Surgery lasted less then 20 minutes | 1 | 0 | 0
Not completed — Entropy failed to detect more than 50% | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 8 | 22 | 18 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 22 | 18 | 48
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 6.63 (3.7) | 24.95 (8.0) | 82.22 (33.8) | 43.38 (37.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 9 | 21
  Male | 4 | 14 | 9 | 27
Region of Enrollment [Number; unit: participants]
  Italy | 8 | 22 | 18 | 48

OUTCOME MEASURES:

1. Primary Outcome: BISPECTRAL Index
Description: The collected values of bispectral index and end tidal sevofluorane will generate a single prediction probability (PK) of agreement between bispectral index vs end-tidal sevofluorane along the whole period of anesthesia for each arm/group.
  Prediction probability (PK) is a statistical measure that is particularly suited to assess the performance of anesthetic depth indicators. It quantifies the correlation between observed anesthetic depth and indicator values. PK allows a simple interpretation and, as a non parametric measure, it is independent from scale units and assumptions on underlying distributions.
Time Frame: BISPECTRAL index values from the induction moment to the awakening moment, 1/5 sec sampling rate, an average of 1 hours
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 8 | 22 | 18
units on a scale | 0.6 [0.57 to 0.61] | 0.66 [0.64 to 0.67] | 0.73 [0.71 to 0.74]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority or Other; p < 0.01, bootstrap

2. Primary Outcome: Entropy
Description: The collected values of Entropy will generate a single prediction probability (PK) of agreement between Entropy vs end-tidal sevofluorane along the whole period of anesthesia for each arm/group.
  Prediction probability (PK) is a statistical measure that is particularly suited to assess the performance of anesthetic depth indicators. It quantifies the correlation between observed anesthetic depth and indicator values. PK allows a simple interpretation and, as a non parametric measure, it is independent from scale units and assumptions on underlying distributions.
Time Frame: Entropy values from the induction moment to the awakening moment, 1/5 sec sampling rate, an average of 1 hours
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 8 | 22 | 18
units on a scale | 0.64 [0.62 to 0.65] | 0.66 [0.65 to 0.68] | 0.72 [0.71 to 0.74]
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Superiority or Other; p < 0.01, bootstrap

3. Secondary Outcome: BISPECTRAL Index Awaking
Description: In each patient the Bispectral index values at the moment of first signs of awakening.The Bispectral index monitor provides a single dimensionless number, which ranges from 0 (equivalent to EEG silence) to 100 (deepest/highest level of anesthesia). A BIS value between 40 and 60 indicates an appropriate level for general anesthesia, as recommended by the manufacturer
Time Frame: reported moment of awakening from anesthesia, an average of 1 hours after administration of Anesthesia
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 8 | 22 | 18
units on a scale | 75 [62 to 78] | 86 [77 to 92] | 81 [74 to 88]
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Entropy Awaking
Description: In each patient the Entropy values at the moment of first signs of awakening. The Entropy monitor provides a single dimensionless number, which ranges from 0 (equivalent to EEG silence) to 100 (deepest/highest level of anesthesia). A Entropy value between 40 and 60 indicates an appropriate level for general anesthesia, as recommended by the manufacturer
Time Frame: reported moment of awakening from anesthesia, an average of 1 hours after administration of Anesthesia
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 8 | 22 | 18
units on a scale | 63 [49 to 71] | 96 [93 to 98] | 86 [78 to 96]
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Whole period of study from January 2014 to November 2014
Description: No adverse events were expected. No adverse events were reported.
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/8 | 0/22 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No